CLINICAL TRIAL: NCT01439958
Title: A Long-term Safety Follow-up Study of L-CsA Therapy for Patients Who Participated in Study 12011.201 and Volunteered to Continue or to Cross-over to L-CsA Inhalation Therapy
Brief Title: Long-term Safety Follow-up Study in the Prevention of Bronchiolitis Obliterans Syndrome (BOS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Core study 12011.201 was terminated.
Sponsor: Pari Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12011.203; 2011-004304-38 (EudraCT Number)
Record Dates: First submitted 2011-09-22; First posted 2011-09-23 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Bronchiolitis Obliterans
Keywords: Inhalation; Lung Transplantation; Cyclosporine
MeSH Terms: conditions — Bronchiolitis Obliterans; Respiratory Aspiration | interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L-CsA (Experimental): Twice daily inhalation of L-CsA
  Interventions: Drug: Inhalation

INTERVENTIONS:
Drug: Inhalation — Twice daily inhalation for a maximum of three years.
  Other Names: aerosolized liposomal CsA

SUMMARY:
The purpose of this study is to evaluate long-term safety of L-CsA in prevention of bronchiolitis obliterans syndrome (BOS) following lung transplantation (LTx) in patients previously enrolled in phase II/III L-CsA clinical trial 12011.201.

DETAILED DESCRIPTION:
This is an uncontrolled extension study open only to patients who completed the Phase II/III core study 12011.201 and volunteered to continue or to cross-over to L-CsA inhalation therapy.

Determination of long-term safety and efficacy outcome over a maximum of three years will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has completed the L-CsA clinical trial 12011.201
2. Patient is capable of understanding the purpose and risks of the follow-up study, has been fully informed and has given written informed consent to participate in the study
3. Female patients of child bearing potential must test negative on standard urine pregnancy test prior to continuation and must agree to practice effective birth control during the study
4. Estimated life expectancy > 6 months
5. Capable of self-administration of medications
6. Patient has stable creatinine levels

Exclusion Criteria:

1. Patients with ongoing irreversible L-CsA related serious adverse events
2. Patients with known hypersensitivity for ciclosporin A
3. Patient intends to participate in another IMP clinical trial other than listed in the inclusion criteria
4. Patient receives mechanical ventilation
5. Patients underwent pulmonary re-transplantation
6. Patient is a pregnant or breast-feeding woman
7. Patient is unlikely to comply with visits, inhalation procedures or spirometric measurements scheduled in the protocol
8. Patient receives any systemic or topical Rosuvastatin
9. Patient has been previously enrolled in this study
10. Patient with malignancy diagnosed during study 12011.201 (with the exception of skin cancer)
11. Documented respiratory infections unless on appropriate antimicrobial therapy with evidence of clinical response
12. Patient is not eligible to continue IMP inhalation according to the Investigator's discretion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Long-term safety of L-CsA in prevention of bronchiolitis obliterans syndrome (BOS) | 3 years
  Safety will be assesses by the numbers of treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) and overall rate of mortality.

SECONDARY OUTCOMES:
Long-term efficacy outcome over a maximum of three years of patients previously enrolled in phase II/III L-CsA clinical trial 12011.201 | 3 years
  Efficacy will be assessed mainly for the following efficacy endpoints:
  * BOS-free survival
  * Incidence of BOS
  * Pulmonary function

CONTACTS AND LOCATIONS:
Overall Officials: Claus Neurohr, MD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- PARI Pharma GmbH, Gräfelfing, Germany